CLINICAL TRIAL: NCT00566371
Title: The Effect of a Once Daily Dose of Atomoxetine (ATX) on ADHD-Related Insomnia
Brief Title: The Effect of a Once Daily Dose of Atomoxetine (ATX) on ADHD-Related Insomnia in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Judith Owens, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 701-1315; 0120-05
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2007-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; Insomnia
Keywords: attention deficit hyperactivity disorder; insomnia; atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients will then be randomized (at Visit 2) to receive either atomoxetine or placebo for 4 weeks (Treatment Period); study drug will be titrated individually according to tolerability and efficacy (measured by ADHD-RS and CGI-I) completed at Visits 3, 4, 5, and 6) at 7-10 day intervals to a maximum dose of 1.8 mg/kg.
  Interventions: Drug: atomoxetine
- 2 (Placebo Comparator): Patients will then be randomized (at Visit 2) to receive either atomoxetine or placebo for 4 weeks (Treatment Period); study drug will be titrated individually according to tolerability and efficacy (measured by ADHD-RS and CGI-I) completed at Visits 3, 4, 5, and 6) at 7-10 day intervals to a maximum dose of 1.8 mg/kg.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine — Patients will then be randomized (at Visit 2) to receive either atomoxetine or placebo for 4 weeks (Treatment Period); study drug will be titrated individually according to tolerability and efficacy (measured by ADHD-RS and CGI-I) completed at Visits 3, 4, 5, and 6) at 7-10 day intervals to a maximum dose of 1.8 mg/kg.
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This study is a single site, double-blind, randomized, placebo-controlled parallel group design. this study is designed to directly examine the efficacy of a single daily dose of atomoxetine taken in the morning in alleviating sleep initiation insomnia in children with ADHD. Primary outcome measures are sleep parameters, specifically mean sleep onset latency (time of onset to persistent sleep), as measured by actigraphy/sleep diary, and parent and child-reported evening settling difficulties, as measured on the evening subscale items of the parent and child versions of the DPREMB-R. Secondary outcome measures include: additional actigraphic sleep parameters (night wakings, sleep duration, and sleep efficiency), daytime sleepiness (Pediatric Daytime Sleepiness Scale, sleepiness visual analogue scale (VAS), and morning behaviors on the DPREMB-R); ADHD symptom improvement (ADHD-RS, parent version; provider-completed CGI); a neurocognitive measure of attention and impulsivity (CPT); executive functions (Brown ADD Scale for Children) and functional outcomes/quality of life (CHQ).

ELIGIBILITY:
Inclusion Criteria:

Subjects are children aged 6 through 17 years with DSM-IV criteria-defined ADHD and sleep initiation insomnia.

Exclusion Criteria:

the sleep onset delay must not be exclusively related to direct or rebound effects of psychostimulant treatment. All subjects will be screened for primary sleep disorders with survey questionnaires (Children's Sleep Habits Questionnaire, CSHQ (12) and Restless Sleep Questionnaire) (Visit 1); subjects scoring above a pre-defined threshold for OSA and/or RLS/PLMD symptoms will be excluded from the study. Other exclusion criteria include IQ < 80 (WISC-III screen at baseline), history of significant chronic medical illness (diabetes, severe asthma), co-morbid depression or other significant psychiatric co-morbidities (ODD, LD not excluded; determined by screening with the Diagnostic Interview Schedule for Children (DISC)), history of chronic use of sedating (eg, antihistamines) or alertness-enhancing (eg, caffeine) medications, history of conditions for which use of atomoxetine is contraindicated (eg, narrow angle glaucoma), use of other prescription medication for ADHD and/or use of prescription/OTC medication for sleep (eg, alpha agonists, hypnotics, melatonin, antihistamines) following the screening visit, and history of failure to respond to an adequate (defined as appropriate dose and adequate duration of therapy) previous trial of atomoxetine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures are sleep parameters, specifically mean sleep onset latency as measured by actigraphy/sleep diary, and parent and child-reported evening settling difficulties. | 3 years

SECONDARY OUTCOMES:
Secondary outcome measures include: additional actigraphic sleep parameters daytime sleepiness, ADHD symptom improvement; a neurocognitive measure of attention and impulsivity, executive functions, and functional outcomes/quality of life. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith Owens, MD, Principal Investigator — Lifespan
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States